CLINICAL TRIAL: NCT02593019
Title: Phase II, Single-arm Study of AZD1775 Monotherapy in Relapsed Small Cell Lung Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Keunchil Park, MD,PhD,Division of hematology-oncology,Department of medicine, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-10-178
Record Dates: First submitted 2015-10-28; First posted 2015-10-30 (Estimated); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — adavosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD1775 (Experimental): AZD1775 175 mg BID per os every 12 hours (6 doses) administered days 1-3 the first week and then days 1-3 the 2nd week of 21 day cycle.
  Interventions: Drug: AZD1775

INTERVENTIONS:
Drug: AZD1775 — AZD1775 175 mg BID per os every 12 hours (6 doses) administered days 1-3 the first week and then days 1-3 the 2nd week of 21 day cycle.
  Tumour evaluation using RECIST 1.1 will be conducted at screening (within 28 days prior to first dose) and every 6 weeks relative to the date of first dose, up to week 42, then every 9 weeks until objective disease progression (within a window of +/- 7 days of the scheduled date).

SUMMARY:
AZD1775 (previously known as MK-1775 in earlier studies) is an inhibitor of Wee1, a protein tyrosine kinase. Wee1 phosphorylates and inhibits cyclin-dependent kinases 1 (CDK1) and 2 (CDK2), and is involved in regulation of the intra-S and G2 cell cycle checkpoints.

CDK1 (also called cell division cycle 2, or CDC2) activity drives a cell from the G2 phase of the cell cycle into mitosis. In response to DNA damage, Wee1 inhibits CDK1 to prevent the cell from dividing until the damaged DNA is repaired (G2 checkpoint arrest).

Inhibition of Wee1 is expected to release a tumor cell from chemotherapeutically-induced arrest of cell replication. In vitro experiments demonstrate that AZD1775 has synergistic cytotoxic effects when administered in combination with various DNA damaging agents that have divergent mechanisms of action. Therefore, the primary objective of the clinical development of AZD1775 is its use as a chemosensitizing drug in combination with a cytotoxic agent (or combination of agents) for treatment of advanced solid tumors.

CDK2 activity drives a cell into, and through, S-phase of the cell cycle where the genome is duplicated in preparation for cell division. Inhibition of Wee1 is expected to cause aberrantly high CDK2 activity in S-phase cells which, in turn, leads to unstable DNA replication structures and ultimately DNA damage. Therefore, it is anticipated that AZD1775 will have independent anti-tumor activity in the absence of added chemotherapy.

The tumor suppressor protein p53 regulates the G1 checkpoint. As the majority of human cancers harbor abnormalities in this pathway they become more dependent on S- and G2- phase checkpoints. Thus, S- and G2-checkpoint abrogation caused by inhibition of Wee1 may selectively sensitize p53-deficient cells.

One hundred percent of Small cell lung cancer has TP53 mutation, therefore we can expect that most of Small cell lung cancer have lost G1 checkpoint and has high probability of WEE1 dependency for proper DNA repair and cell cycle progression. For this reason, Small cell lung cancer could be a good clinical trial target disease for WEE1 inhibitor.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of fully informed consent prior to any study specific procedures.
2. Patients must be ≥20 years of age.
3. Small cell lung cancer that has progressed during or after first-line therapy.

   * The 1st line regimen must have contained platinum based regimen.
   * Refractory to first-line chemotherapy or relapse within 6 months since the last dose of first-line chemotherapy
   * If the patient correspond to sensitive relapse (relapse more than 6 months since the last dose of first-line chemotherapy), she/he should get second-line treatment.
4. Previous radiotherapy is allowed.
5. Provision of tumor sample (from either archival or fresh biopsy)
6. Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
7. ECOG performance status 0-2
8. Patients must have a life expectancy ≥ 3 months from proposed first dose date.
9. Patients must have acceptable bone marrow, liver and renal function measured within 14 days prior to administration of study treatment as defined below:

   * Haemoglobin ≥9.0 g/dL
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * White blood cells (WBC) > 3 x 109/L
   * Platelet count ≥100 x 109/L - Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
   * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case it must be ≤ 5x ULN
   * Serum creatinine ≤1.5 x institutional ULN and a calculated creatinine clearance (CrCl) ≥45 mL/min by the Cockcroft-gault method:

   CrCl = (140-age) x (weight/kg) x (0.85 if female) (72 x serum creatinine mg/dL)
10. At least one measurable lesion that can be accurately assessed by imaging or physical examination at baseline and follow up visits.
11. Negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on day 1, if woman of childbearing potential
12. Female patients who are not of childbearing potential and fertile female patients of childbearing potential who agree to use adequate contraceptive measures, who are not breastfeeding.
13. Fertile male patients willing to use at least one medically acceptable form of birth control, and must not donate sperm, for the duration of the study, and for 2 weeks after treatment stops

Exclusion Criteria:

1. More than two prior chemotherapy regimen for the treatment of small cell lung cancer
2. Any previous treatment with P53 inhibitors (small molecules)
3. Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for >2 years.
4. Patients unable to swallow orally administered medication.
5. Treatment with any investigational product during the last 14 days before the enrollment (or a longer period depending on the defined characteristics of the agents used).
6. Patients receiving any systemic chemotherapy, radiotherapy (except for palliative reasons), within 3 weeks from the last dose prior to study treatment (or a longer period depending on the defined characteristics of the agents used). The patient can receive a stable dose of bisphosphonates or denosumab for bone metastases, before and during the study as long as these were started at least 4 weeks prior to treatment.
7. Concomitant use of known sensitive CYP3A4 substrates or CYP3A4 substrates with a narrow therapeutic index, or to be moderate to strong CYP3A4 inhibitor/inducer which cannot be discontinued to weeks prior to Day 1 of dosing and withheld throughout the study until 2 weeks after the last dose of study drug, Co-administration of aprepitant or fosaprepitant during this study is prohibitedRefer to the Section 5.9.2 and Appendix H for listing of all prohibited medications.
8. With the exception of alopecia, any ongoing toxicities (>CTCAE grade 1) caused by previous cancer therapy.
9. Intestinal obstruction or CTCAE grade 3 or grade 4 upper GI bleeding within 4 weeks before the enrollment.
10. Resting ECG with measurable QTcB > 480 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.
11. Patients with cardiac problem as follows: unstable angina pectoris, congestive heart failure, acute myocardial infarction, conduction abnormality not controlled with pacemaker or medication, significant ventricular or supraventricular arrhythmias (patients with chronic rate controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible).
12. Female patients who are breast-feeding or child-bearing
13. Any evidence of severe or uncontrolled systemic disease, active infection, active bleeding diatheses or renal transplant, including any patient known to have human immunodeficiency virus (HIV), active hepatitis B or active hepatitis C
14. Major surgical procedures ≤28 days of beginning study treatment, or minor surgical procedures ≤7 days
15. Known central nervous system (CNS) disease other than neurologically stable,treated brain metastases - defined as metastasis having no evidence of progression or haemorrhage for at least 2 weeks after treatment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-12; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Objective reponse rate | Up to 24 weeks for each subject

SECONDARY OUTCOMES:
Duration of response | Up to 24 weeks for each subject
Disease control rate | 8 weeks
Overall survival (OS) | Up to 24 weeks for each subject
progression-free survival (PFS) | Up to 24 months for each subject
Number of subjects with Adverse Events as a Measure of Safety and Tolerability | Up to 24 months for each subject

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea